CLINICAL TRIAL: NCT01822704
Title: Application of Vertical Whole Body Vibration in Stroke Patients: Neuromuscular Effects, and Clinical Efficacy
Brief Title: Whole Body Vibration in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20130209001
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Rehabilitation; Vibration
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): This group will undergo three 45-minute exercise sessions per week for 10 weeks. No whole body vibration will be given.
  Interventions: Behavioral: Leg exercises
- Low intensity vibration (Experimental): This group will receive three 45-minute whole body vibration training sessions for 10 consecutive weeks. The vibration will be of low intensity (frequency: 20 Hertz, amplitude: 1mm).
  Interventions: Device: Low intensity whole body vibration; Behavioral: Leg exercises
- High intensity vibration (Experimental): This group will receive three 45-minute whole body vibration training sessions per week for 10 consecutive weeks.The vibration will be of higher intensity than the low intensity vibration group (frequency: 30 Hertz, amplitude: 1mm).
  Interventions: Device: High intensity whole body vibration; Behavioral: Leg exercises

INTERVENTIONS:
Device: Low intensity whole body vibration
  Arms: Low intensity vibration
Device: High intensity whole body vibration
  Arms: High intensity vibration
Behavioral: Leg exercises

SUMMARY:
This study is a randomized controlled trial aimed to assess the efficacy of a 10-week whole body vibration training program on physical functioning, societal participation and quality of life in individuals with chronic stroke. It is hypothesized that the whole body vibration program will induce significantly more gain in physical functioning, societal participation, and quality of life in chronic stroke patients, compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a hemispheric stroke
* chronic stroke (onset of 6 months or more)
* aged 18 years or older
* medically stable
* able to stand for at least 1 minute with hand support
* Abbreviated Mental Test score at 6 or more
* Chedoke McMaster Stroke Assessment leg or foot score less than 7 points

Exclusion Criteria:

* recurrent stroke
* brainstem or cerebellar stroke
* other neurological conditions
* significant musculoskeletal conditions (e.g. amputations)
* vestibular disorders
* peripheral vascular disease
* other serious illnesses
* other contraindications to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-11 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Isometric knee muscle strength | Week 0
Isometric knee muscle strength | week 10

SECONDARY OUTCOMES:
Eccentric knee muscle strength at a velocity of 60 degrees per second | Week 0
Eccentric knee muscle strength at a velocity of 60 degrees per second | week 10
Concentric knee muscle strength at a velocity of 60 degrees per second | week 0
Concentric knee muscle strength at a velocity of 60 degrees per second | week 10
Distance walked in the Six Minute Walk Test | week 0
Distance walked in the Six Minute Walk Test | week 10
Average oxygen consumption rate during the Six Minute Walk Test | week 0
Average oxygen consumption rate during the Six Minute Walk Test | week 10
Time taken to complete the Timed Up and Go Test | week 0
Time taken to complete the Timed Up and Go Test | week 10
Time taken to complete the Five-times-sit-to-stand test | week 0
Time taken to complete the Five-times-sit-to-stand test | week 10
Distance reached in the Functional Reach test | Week 0
Distance reached in the Functional Reach test | week 10
Balance score as measured by the Mini-Balance Evaluation Systems Test | week 0
Balance score as measured by the Mini-Balance Evaluation Systems Test | week 10
Walking ability as measured by the Functional Ambulation Category | week 0
Walking ability as measured by the Functional Ambulation Category | week 10
Balance confidence scores as measured by the Activities-specific Balance Confidence Scale | week 0
Balance confidence scores as measured by the Activities-specific Balance Confidence Scale | week 10
Quality of life score as measured by the 12-item Short Form Health Survey | week 0
Quality of life score as measured by the 12-item Short Form Health Survey | week 10
Level of activity participation as measured by the Frenchay Activities Index | week 0
Level of activity participation as measured by the Frenchay Activities Index | Week 10
Level of perceived environmental barriers as measured by the Craig Hospital Inventory of Environmental Factors | week 0
Level of perceived environmental barriers as measured by the Craig Hospital Inventory of Environmental Factors | week 10
Ankle spasticity score as measured by the Modified Ashworth Scale | week 0
Ankle spasticity score as measured by the Modified Ashworth Scale | week 10

CONTACTS AND LOCATIONS:
Overall Officials: Marco YC Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

REFERENCES:
- [Background] Lau RW, Yip SP, Pang MY. Whole-body vibration has no effect on neuromotor function and falls in chronic stroke. Med Sci Sports Exerc. 2012 Aug;44(8):1409-18. doi: 10.1249/MSS.0b013e31824e4f8c. PMID 22330025